CLINICAL TRIAL: NCT01584414
Title: Evaluation of the Zetiq Histological and Cytological Staining Technique for the Detection Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, fishman ami, Ami Fishman, Meir Medical Center
Other Study IDs: ZT-CL-01A
Record Dates: First submitted 2012-04-22; First posted 2012-04-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Cervical Cancer
Keywords: Zetiq CellDetect ® stain; distinct red/purple color to the cytoplasm of neoplastic; distinguishes green/blue stained non-neoplastic cells and tissues
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- normal samples
- premalignant/carcinoma samples

SUMMARY:
Zetiq has introduced a histochemical stain that claims to tinctorially identify cancer and neoplastic cells. Because of the potential importance of such a capability, the investigators undertook to investigate Zetiq's CellDetect® staining technology as applied to cultured cell lines as well as an initial sample of clinical cases. This goal was pursued by investigating four types of comparisons: 1) cancer cell lines before and after differentiation; 2) cervical squamous-cell carcinoma (SCC) biopsies to non-neoplastic squamous epithelium; 3) SCCs to neoplastic, nonmalignant squamous epithelium; and 4) neoplastic squamous cells to non-neoplastic squamous cells in cytological preparations. The clinical material was also stained with hematoxylin and eosin (biopsies) or Pap (cytologies) for diagnostic purposes. The investigators found that all CellDetect®-stained cells exhibited one of the two tinctorial outcomes. Cell lines with malignant phenotype uniformly had red/purple cytoplasm, whereas the differentiated phenotype changed the color to blue/green.

ELIGIBILITY:
Inclusion Criteria:

1. FEMALE SUBJECT BETWEEN 18 AND 75 YEARS OF AGE.
2. ABILITY TO PROVIDE INFORMED CONSENT

Exclusion Criteria:

1. SUBJECT WITH KNOWN PREGNANCY AT TIME OF SCREENING.
2. PREVIOUS HISTORY OF HYSTERECTOMY
3. PARTICIPATION IN ANOTHER CLINICAL TRIAL WITHIN LAST 30 DAYS.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 archival cervical biopsy cases with the following diagnoses: normal, 22 cases; CIN-2/3, 18 cases; squamous cell carcinoma, 20 cases.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2007-10; Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ami Fishman, Prof, Principal Investigator — Meir medical Center, affiliated with Sackler School of Medicine, Tel-Aviv University
Locations (1):
- Meir Medical Center, Kfar Saba, Israel